CLINICAL TRIAL: NCT07101107
Title: Socio-cognitive and Biological Responses to Childhood Maltreatment in Individuals With Bipolar Disorder and Control Subjects
Brief Title: Socio-cognitive and Biological Responses to Maltreatment
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Collaborators: Medical School Hamburg (Other); University of Innsbruck (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1410/2020; 10.55776/KLP7245424 (Other Grant/Funding Number: The Austrian Science Fund (FWF))
Record Dates: First submitted 2025-07-10; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Bipolar 1 Disorder; Control Subjects
Keywords: childhood maltreatment; Social Cognition; empathy; Bipolar Disorder; Biomolecules; Magnetic Resonance Imaging; Theory Of Mind; telomere length; mitochondria
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells (PBMC), plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bipolar 1 disorder
- Control subjects

SUMMARY:
The study will investigate how a history of emotional childhood maltreatment (CM) is associated with different aspects of psychological (social behaviour, empathy) and biological (brain function and structure, inflammation) health. In fact, CM is a risk factor for many mental disorders, such as schizophrenia and autism. However, it is unclear how a history of emotional CM affects psychological and biological outcomes in bipolar disorder (BD). Therefore, this study focuses on understanding how a possible history of CM affects BD compared to control participants (CP) with no known psychiatric illness.

The aim of the project is to investigate how a history of emotional CM is associated with social cognition. The investigators will recruit 80 CP and 80 people diagnosed with BD, some of whom will have a history of CM. The investigators will assess psychological well-being (social behaviour, empathy) at two points in time at the Department of Psychiatry, Psychotherapy, Psychosomatics and Medical Psychology at the Medical University of Innsbruck (MUI). Additionally, as they want to understand how emotional CM affects brain function and structure, the investigators will perform magnetic resonance imaging (MRI) of the brain at the Neuroimaging Core Facility (Medical University of Innsbruck). The investigators also want to understand how biological markers in the blood (such as telomere length, inflammation) might be affected, assessed in collaboration with the Department of Psychology (Leopold-Franzens University of Innsbruck). Finally, the investigators will look at a combination of the psychological and biological tests to see if there is a link between emotional CM and health outcomes.

DETAILED DESCRIPTION:
Although the contribution of childhood maltreatment (CM) to psychological (e.g. social cognition) and biological (e.g. neural, biomolecular) outcomes has been extensively studied, e.g. in schizophrenia and autism, its contribution to bipolar disorder (BD) and the role of different CM subtypes, multiplicity and timing remains unclear. The aim of the project is to investigate how a history of emotional CM is associated with multidimensional aspects of social cognitive, neural and biomolecular parameters.

The research questions addressed in this project are: i) How is a history of emotional CM associated with social cognition in control participants (CP) with no known psychiatric illness and in individuals diagnosed with BD? ii) How is a history of emotional CM related to biomolecular and neural parameters in CP and individuals diagnosed with BD? iii) How are biomolecular markers, neural parameters, and social cognitive skills related in individuals with a history of emotional CM? The primary aim of this study is to investigate the association of self-reported history of emotional CM with social cognition (i.e. emotion recognition, cognitive and affective empathy) in CP and in individuals diagnosed with BD, both with and without a history of CM. Additional aims are to characterize the association of history of emotional CM with neural (i.e. task-based and resting-state functional magnetic resonance imaging (rs-fMRI), morphometry, white matter) MRI parameters and biomolecular markers (i.e. telomere length, mitochondrial bioenergetics and biogenesis) in peripheral blood mononuclear cells and blood plasma (selected immune-response mediators).

Recruitment, clinical assessments (e.g. Maltreatment and Abuse Chronology of Exposure scale) and blood sampling of 80 CP and 80 individuals diagnosed with BD with and without a history of CM will be performed at two timepoints at the Department of Psychiatry, Psychotherapy, Psychosomatics and Medical Psychology, Medical University of Innsbruck (MUI). Longitudinal MRI acquisitions will be performed at the Neuroimaging Core Facility (MUI). Clinical, MRI and biomolecular analyses will be applied, and correlations of these findings with emotional CM, multiplicity and timing will be evaluated.

The contribution of a history of emotional CM to psychological and biological outcomes in BD is unknown. This study will clarify the association between emotional CM and social cognition in BD and CP. It will study how emotional CM alters brain function and structure in regions related to social cognition. A translational approach combining MR neuroimaging with psychoneuroimmunological methods will assess neural parameters together with biomolecular markers from whole blood in relation to emotional CM and social cognition.

ELIGIBILITY:
Inclusion Criteria for individuals diagnosed with bipolar disorder (BD):

* diagnosis of a moderate to severe depressive episode without psychotic features in the context of BD-I according to the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5: 296.52 BD-I, most recent episode depressed, moderate; 296.53 BD-I, most recent episode depressed, severe without psychotic features;
* Montgomery-Åsberg Depression Rating Scale (MADRS) score≥20;
* age between 18 and 65 years; and
* able to provide written informed consent for magnetic resonance imaging (MRI) and study participation.

Exclusion Criteria for individuals diagnosed with BD:

* a history of one or more diagnoses of the following DSM-5 categories: past or current moderate or severe substance dependence (303.x, 304.x, 305.x) with the exclusion of tobacco use disorder (305.1), neurodevelopmental disorders (299.x, 307.x, 314.x, 315.x, 319.x), schizophrenia spectrum and other psychotic disorders (293.x, 295.x, 297.x, 298.x), neurocognitive disorders (290.x, 292.x, 294.x, 331.x), BD-I Single Manic (296.0x), BD-I Manic (296.4x), BD-I Mixed (296.6, 296.7, 296.8, 296.9), BD-II (296.89), or comorbid Borderline Personality Disorder (BPD) as assessed by Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-PD);
* a current episode of illness with psychotic features (296.54);
* a recent history of central nervous system (CNS) trauma or significant CNS trauma;
* physical illness that might interfere with the participant's cognitive performance;
* an autoimmune disorder or inflammatory diseases;
* currently on anti-inflammatory drugs, cortisol or cortisol derivates;
* cardiovascular impairment with life-threatening issues;
* electroconvulsive therapy in the last 12 months;
* current substance abuse (except caffeine and nicotine) as assessed by DSM-5 or positive urine drug screen;
* IQ≤70 as assessed by the Mehrfachwahl-Wortschatztest" version B (MWT-B);
* MRI contraindications (e.g. claustrophobia, metal, electric, magnetic or mechanically driven implants); or
* other ethical considerations (e.g. pregnancy, lactation, participants not fluent in the language of the cognitive batteries and questionnaires).

Inclusion Criteria for healthy volunteers:

* absence of any axis I disorder according to DSM-5 and physical illness that might interfere with participant's cognitive performance;
* age between 18 and 65 years according to clinical group; and
* ability to give written informed consent for MRI and study participation.

Exclusion Criteria for healthy volunteers:

* first degree relatives with BD, schizophrenia, or known genetically-based mitochondriopathies;
* a history of any axis I disorder, neurological, developmental disorders, CNS trauma, or comorbid BPD.
* physical illness that might interfere with the participants' cognitive performance;
* an autoimmune disorder or inflammatory diseases;
* currently on anti-inflammatory drugs, cortisol or cortisol-derivates;
* cardiovascular impairments with life-threatening issues;
* current substance abuse;
* IQ≤70;
* MRI contraindications; or
* other ethical considerations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For bipolar disorder with a current diagnosis of depressive episode: Inpatient clinic of the Department of Psychiatry, Psychotherapy, Psychosomatics and Medical Psychology of the Medical University Innsbruck.
  For healthy controls: recruitment is done via public advertisements (e.g. posters, flyers, local newspaper announcements) and at the homepage of Medical University Innsbruck, Tirol Kliniken, and University of Innsbruck.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure; MACE-X) and emotion recognition of adult faces (Reading the Mind in the Eyes Test; RMET) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (as assessed by a combined score of the Maltreatment and Abuse Chronology of Exposure [MACE-X] emotional subscales: parental verbal abuse, parental nonverbal emotional abuse, emotional neglect, peer verbal abuse) and emotion recognition (number of correctly identified emotions) as assessed by the Reading the Mind in the Eyes Test adult version (RMET). RMET use expressions from images of 28 adult faces, 50% male and 50% female. The task consist of two types of trials: emotion recognition and sex judgment. In the emotion recognition trials, participants select among four adjectives the one that best describes what the person in the image is thinking or feeling. This task is sensitive to subtle emotion processing deficits since it involves the recognition of a relatively wide range of complex mental states.
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and emotion recognition of child faces (Reading the Mind in the Eyes Test; RME-C-T) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and emotion recognition (number of correctly identified emotions) as assessed the Reading the Mind in the Eyes Test child version (RME-C-T). RME-C-T uses high-quality pictures of 28 child faces. The task consist of two types of trials: emotion recognition and sex judgment. In the emotion recognition trials, participants select among four adjectives the one that best describes what the person in the image is thinking or feeling.
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and cognitive empathy (Multifaceted Empathy Test; MET-core 2) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and cognitive empathy (number of correctly identified) as assessed by The Multifaceted Empathy Test (MET-core 2). MET-core 2 is an ecologically valid measure that allows separate assessment of cognitive and affective empathy. It consists of 40 photographs depicting people in emotionally charged situations and is designed to elicit strong emotional reactions. To assess cognitive empathy ("What is the person feeling?"), the mental states of the people in the photographs are selected from four mental state descriptors. To assess affective empathy ("How much are you feeling for the person?"), the level of empathic concern for the depicted individuals is rated on a 4-point Likert scale (from "not at all" to "very strong") for the same series of pictures.
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and affective empathy (Multifaceted Empathy Test; MET-core 2) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and affective empathy (rating) as assessed by The Multifaceted Empathy Test (MET-core 2). MET-core 2 is an ecologically valid measure that allows separate assessment of cognitive and affective empathy. It consists of 40 photographs depicting people in emotionally charged situations and is designed to elicit strong emotional reactions. To assess cognitive empathy ("What is the person feeling?"), the mental states of the people in the photographs are selected from four mental state descriptors. To assess affective empathy ("How much are you feeling for the person?"), the level of empathic concern for the depicted individuals is rated on a 4-point Likert scale for the same series of pictures.

SECONDARY OUTCOMES:
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and brain morphometry (T1-weighted imaging) | At enrollment (bipolar disorder with moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and brain morphometry (T1-weighted MRI). The research hypothesis is that increasing severity of a history of emotional childhood maltreatment will correlate with small limbic volumes (e.g. hippocampi, amygdala, thalamus). These changes in morphometry will be more pronounced in bipolar disorder compared to control participants.
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and brain responses (task-based fMRI) | At enrollment (bipolar disorder with moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and brain responses (task-based functional MRI). In control participant, the hypothesis is that increasing severity of a history of emotional childhood maltreatment will correlate with: i) low brain responses during RMET/RME-C-T (along with correct and rapid identification of negative emotions) in social cognitive brain regions (e.g. temporoparietal junction, medial prefrontal cortex, amygdala, insula); ii) high brain responses during MET-Core 2 (along with high cognitive and affective empathy abilities). In bipolard disorder, increasing severity of a history of emotional childhood maltreatment will correlate with: i) high brain responses during RMET/RME-C-T in social cognitive regions (along with incorrect and slow identification of negative emotions) ii) low brain responses during MET-Core 2 (along with low cognitive and affective empathy abilities).
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and brain functional connectivity (resting-state functional MRI). | At enrollment (bipolar disorder with moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and brain functional connectivity (resting-state functional MRI). The hypothesis is that increasing severity of a history of emotional childhood maltreatment will correlate low functional connectivity within the Theory-of-Mind (ToM) network. These changes in functional connectivity will be more pronounced in bipolar disorder compared to control participants. Both cognitive and affective ToM tasks involve the posterior temporoparietal junction, the posterior superior temporal sulcus, and the posterior cingulate cortex. While cognitive ToM involves the dorsolateral prefrontal cortex (PFC), dorsal striatum, dorsal anterior cingulate cortex (ACC), and dorsomedial PFC, affective ToM involves the inferior frontal gyrus, insula, ventral striatum, amygdala, temporal poles, ACC, and medial PFC.
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and brain white matter values (diffusion MRI) | At enrollment (bipolar disorder with moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and brain white matter values (diffusion MRI). The hypothesis is that increasing severity of a history of emotional childhood maltreatment will correlate with disruption (e.g. low fractional anisotropy values) in white matter tracts connecting social cognitive regions (e.g. superior longitudinal fasciculus, cingulum, uncinate fasciculus, corpus callosum). These changes in white matter will be more pronounced in bipolar disorder compared to control participants.
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and inflammation | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and inflammation (measured from blood samples). The hypothesis is that increasing severity of a history of emotional childhood maltreatment is correlated with higher inflammation levels (e.g. CRP, IL-1β, IL-6, TNF-α). High levels of inflammation will be more pronounced in bipolar disorder compared to control participants.
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and telomere length | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and telomere length (measured from blood samples). The hypothesis is that increasing severity of a history of emotional childhood maltreatment is correlated with telomere shortening. Telomere shortening will be more pronounced in bipolar disorder compared to control participants.
Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and mitochondrial bioenergetics and biogenesis | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  Correlation between a history of emotional childhood maltreatment score (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) and mitochondrial bioenergetics and biogenesis (measured from blood samples). The hypothesis is that in control participants increasing severity of a history of emotional childhood maltreatment is correlated with high mitochondria function (e.g. high mitochondrial respiratory activity and density as a compensatory effect of chronic stress) whereas in bipolar disorder it will correlate with impairments in mitochondria function.

OTHER OUTCOMES:
Illness effects and stability of self-reported childhood maltreatment assessment | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) assessments of self-reported childhood maltreatment (Maltreatment and Abuse Chronology of Exposure scale; MACE-X) data are used to study the illness effects in bipolar disorder and stability of assessments in control participants.
Illness effects and stabilitity of emotion recognition (RME-C-T) | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) assessment of emotion recognition (number of correctly identified emotions) as assessed the Reading the Mind in the Eyes Test child version (RME-C-T) is used to study the illness effects in bipolar disorder and stability of assessments in control participants.
Illness effects and stabilitity of emotion recognition (RMET) | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) assessment of emotion recognition (number of correctly identified emotions) as assessed by the Reading the Mind in the Eyes Test adult version (RMET) is used to study the illness effects in bipolar disorder and stability of assessments in control participants.
Illness effects and stabilitity of cognitive empathy (MET-core 2) | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) assessment of cognitive empathy (number of correctly identified) as assessed by The Multifaceted Empathy Test (MET-core 2) is used to study the illness effects in bipolar disorder and stability of assessments in control participants.
Illness effects and stabilitity of affective empathy (MET-core 2) | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) assessment of affective empathy (rating) as assessed by The Multifaceted Empathy Test (MET-core 2) is used to study the illness effects in bipolar disorder and stability of assessments in control participants.
Illness effects and stability of brain responses (task-based fMRI responses) | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) assessments of brain responses during task-based fMRI (RME-C-T, RMET, MET-core-2) are used to study the illness effects in bipolar disorder and stability of assessments in control participant
Illness effects and stability of brain functional connectivity (resting-state fMRI) | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) assessments of brain functional connectivity (resting-state fMRI) are used to study the illness effects in bipolar disorder and stability of assessments in control participants.
Illness effects and stability of brain white matter values (diffusion MRI) | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) assessments of brain white matter values (diffusion MRI) are used to study the illness effects in bipolar disorder and stability of assessments in control participants.
Illness effects and stability of brain morphometry (T1-weighted imaging) | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) assessments of brain morphometry (T1-weighted imaging) are used to study the illness effects in bipolar disorder and stability of parameters in control participants.
Illness effects and stability of telomere length | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) telomere length (assessed from blood samples) are used to study the illness effects in bipolar disorder and stability of assessments in control participants.
Illness effects and stability of mitochondrial bioenergetics and biogenesis | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) mitochondrial bioenergetics and biogenesis (assessed from blood samples) are used to study the illness effects in bipolar disorder and stability of assessments in control participants.
Illness effects and stability of inflammatory parameters | Between enrollment (depressive) and improved clinical states (remission, response) at 3-6 months after enrollment in bipolar disorder. In control participants, at enrollment and at 3-6 months after.
  Change in the baseline and follow-up (3 to 6 months) of inflammatory (assessed from blood samples) parameters are used to study the illness effects in bipolar disorder and stability of assessments in control participants
Psychological distress with the Mini-Symptom-Checklist (Mini-SCL) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  The Mini-Symptom-Checklist (Mini-SCL) assesses symptomatic stress with 18 questions on a Likert scale ranging from 0 (not at all) to 4 (very strongly). Higher scores on the Mini-SCL indicate higher levels of psychological distress or symptom severity
Brief Assessment of Cognition in Schizophrenia (BACS) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  The Brief Assessment of Cognition in Schizophrenia (BACS) is used to rule out impairment in non-social cognition, i.e. verbal memory, working memory, motor speed, verbal fluency, attention and processing speed, and executive functions. It has high reliability and has been validated in several languages. BACS raw values are converted into T values with a mean of 50 and a standard deviation of 10. In summary, while there isn't a fixed maximum or minimum score, lower BACS scores (especially when below -1 or -2 on the Z-score scale) are indicative of cognitive deficits. The BACS was originally developed for schizophrenia but has been used in individuals diagnosed with bipolar disorder who achieved lower scores in the composite and most subtest scores compared to control participants.
Mini-International Neuropsychiatric Interview (M.I.N.I.) | At screening
  Any Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 psychiatric disorders will be screened with Mini-International Neuropsychiatric Interview (M.I.N.I.) version 7.0.2 on the recruitment stage. The M.I.N.I. is a validated, structured, diagnostic interview tool with high diagnostic reliability, consisting of questions that parallel symptoms in the DSM. M.I.N.I. has 17 modules. Each question within a module is answered with a "yes" or "no". A "yes" answer contributes one point to the module's score. Clinicians sum the positive responses to determine the module score, which indicates whether the participant meets the diagnostic criteria for that particular disorder.
The Montgomery-Åsberg Depression Rating Scale (MADRS) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment.
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item questionnaire used to determine the degree of depressive symptoms in individuals diagnosed with bipolar disorder and subclinical depression in control participants. Each item yields a score ranging from 0 to 6, and the overall score ranges from 0 to 60. Higher MADRS scores indicate more severe depressive symptoms.
German multiple-choice vocabulary test MWT-B | Screening
  IQ is assessed with German multiple-choice vocabulary test (MWT-B). It assesses crystallized intelligence. It consists of 37 items of multiple choice (5 words) vocabulary test. One of the answers is correct. Maximum of 37 correct words corresponds to IQ=120.
Young Mania Rating Scale (YMRS) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment.
  Young Mania Rating Scale (YMRS) assesses the severity of manic symptoms with 11 items. The overall score ranges from 0 to 60 with higher scores indicating more severe mania. Each item is scored either on a 0 to 4 scale (7 items) or with twice the scaling weight from 0 to 8 (4 items).
Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-PD) | Screening
  Comorbid borderline personality disorder is assessed by Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-PD). It is used to assess comorbid borderline personality disorder traits (14 questions) which are often found in an interaction between bipolar disorder and childhood maltreatment. Higher scores indicate a greater severity of personality pathology.
Toronto Alexithymia Scale (TAS) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  The Toronto Alexithymia Scale (TAS) consists of 20 statements on a 5-point Likert scale which measure participants' difficulties in identifying or describing their own emotions (1=strongly disagree/5=strongly agree), and their externally oriented thinking style which allows reliable discrimination of alexithymic and non-alexithymic individuals. The TAS-20 has 3 subscales: Difficulty Describing Feelings, Difficulty Identifying Feeling, and Externally-Oriented Thinking. There are 5 items that are negatively keyed. The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 =possible alexithymia. MET and RMET performance correlates negatively with TAS scores, which is expected as empathetic traits facilitate and alexithymic traits impair emotion recognition.
Interpersonal Reactivity Index (IRI) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  The IRI consists of 28 statements on a 5-point Likert scale (scored from 0 to 4) which requires participants to decide on other-directed thoughts and feelings (Does not describe me well/Describes me very well), and is a widely used multidimensional measure of trait empathy. The measure has 4 subscales, each made up of 7 different items: Perspective taking (PT), Fantasy (FS), Empathic concern (EC), and Personal Distress (PD), where higher scores generally indicate a greater tendency towards empathy. MET and RMET performance correlates positively with IRI, which is expected as empathetic traits facilitate and alexithymic traits impair emotion recognition. EC and PD scales have been referred to as measuring affective empathy while the PT and FS scale are commonly referred to as measuring cognitive empathy.
The resource allocation task (RAT-6) | In bipolar disorder, at enrollment (in moderate or severe depressed state) and at improved clinical state (response or remission) at 3-6 months after enrollment. In control participants, at enrollment and at 3-6 months after.
  The resource allocation task (RAT-6) measures prosociality with 6 decisions regarding the imaginary split of money between the participant and another person, where nine options are given. The set of responses can then be scored to yield a single score, the rank order of social preferences (altruistic, prosocial, individualistic, and competitive), and additionally contains a check for transitivity in revealed preferences. Given the angles that result from idealized SVO types, proper boundaries between categories can be derived by bisecting the respective adjacent ranges. Altruists would have an angle greater than 57.15◦; prosocials would have angles between 22.45◦ and 57.15◦; individualists would have angles between -12.04◦ and 22.45◦ ; and competitive types would have an angle less than -12.04◦. Mindreading performance predicts RAT performance which indicates its real consequences on social behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FWF Austrian science fund website — https://www.fwf.ac.at/forschungsradar/10.55776/KLP7245424
- See also: Reposity to store study results — https://zenodo.org/communities/fwf_10_55776_klp7245424/records?q=&l=list&p=1&s=10&sort=newest